CLINICAL TRIAL: NCT02761863
Title: Effect of Expression of CD74 and VEGF on Outcome of Treatment in Patients With Malignant Pleural Mesothelioma Receiving Pemetrexed/Platinum Protocol
Brief Title: Effect of Expression of CD74 and VEGF on Outcome of Treatment in Patients With Malignant Pleural Mesothelioma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Nagy, Dr, Ain Shams University
Other Study IDs: CURE001
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Mesothelioma; CD 74; VEGF
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paraffin Blocks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CD74 - VEGF arm
  Interventions: Other: CD 74, VEGF detection

INTERVENTIONS:
Other: CD 74, VEGF detection — All MPM samples will be subjected to immunohistochemistry with CD74 and VEGF antibodies.
  The VEGF will be scored using a 0-3 scoring system to represent the percentage of cytoplasmic positively stained cells in the tumor portion, as follows: 0-10%, 11-30%, 31-60% and 61-100% positive staining correspond to score 0, 1, 2 and 3 respectively. Both CD74 and VEGF immunohistochemical markers will be furtherly categorized in the statistical analyses as none (0)/low (1) vs medium (2)/high expression(3).
  The CD74 expression will be recorded in the tumor and the stroma semiquantitatively using the histoscore method using four representative fields with the final score resulting from the percentage of tumor cells staining positively multiplied by the staining intensity grade.

SUMMARY:
This is a prospective study evaluating the effect of expression of CD74 and VEGF on outcome of treatment in patients with malignant pleural mesothelioma receiving Pemetrexed/Platinum protocol. The paraffin blocks of the patients will be tested for CD74 and VEGF before starting treatment using IHC and the results will be correlated with the outcome of treatment during evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of malignant pleural Mesothelioma
2. No prior chemotherapy.
3. ECOG less than or equal to 2 .
4. Measurable disease according to the requirements of SWOG criteria.
5. Age ≥ 19 years .
6. Estimated life expectancy of at least 12 weeks .
7. Adequate bone marrow reserve (white blood cells [WBC] ≥ 3.5 × 109 /L, neutrophils ≥ 1.5 × 109 /L, platelets ≥ 100 × 109 /L, and hemoglobin ≥ 9.0 gm/dL).

Exclusion Criteria:

1. Presence of central nervous system metastases.
2. Inadequate liver function (bilirubin > 1.5 times upper normal limit [UNL] and alanine transaminase [ALT] or aspartate transaminase [AST] > 3.0 UNL or up to 5.0 UNL in the presence of hepatic metastases).
3. Inadequate renal function (creatinine > 1.25 times UNL, creatinine clearance < 50mL/min).
4. Serious concomitant systemic disorder incompatible with the study.
5. Second primary malignancy (except in situ carcinoma of the cervix, adequately treated basal cell carcinoma of the skin, T1 vocal cord cancer in remission, or prior malignancy treated more than 5 years prior to enrollment without recurrence).
6. Pregnancy

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Malignant Pleural Mesothelioma
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-30 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
CD 74 and VEGF detection effect on response to treatment | Essay done before starting treatment and correlated with the response
  The paraffin blocks of the patients will be tested for CD74 and VEGF before starting treatment using IHC and the results will be correlated with the outcome of treatment during evaluation.
  All MPM samples will be subjected to immunohistochemistry with CD74 and VEGF antibodies.
  The VEGF will be scored using a 0-3 scoring system to represent the percentage of cytoplasmic positively stained cells in the tumor portion, as follows: 0-10%, 11-30%, 31-60% and 61-100% positive staining correspond to score 0, 1, 2 and 3 respectively. Both CD74 and VEGF immunohistochemical markers will be furtherly categorized in the statistical analyses as none (0)/low (1) vs medium (2)/high expression(3).
  The CD74 expression will be recorded in the tumor and the stroma semiquantitatively using the histoscore method using four representative fields with the final score resulting from the percentage of tumor cells staining positively multiplied by the staining intensity grade.

IPD SHARING:
Plan to Share IPD: No